CLINICAL TRIAL: NCT02107235
Title: Phase I Study of Platinum-based Chemoradiotherapy (CRT) With Oral Rigosertib in Patients With Intermediate or High-risk Head and Neck Squamous Cell Carcinoma
Brief Title: Platinum-based Chemoradiotherapy and Rigosertib in Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 09-12
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Head and Neck Neoplasms; Carcinoma, Squamous Cell
Keywords: Chemoradiotherapy; cisplatin
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — ON 01910; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rigosertib + Cisplatin + Radiation (Experimental): Oral rigosertib will be started 7 days before initiation of concurrent treatment with cisplatin and radiation therapy and will be administered on a continuous basis for a fixed duration of 8 weeks. Three oral rigosertib escalating doses will be sequentially evaluated: 70 mg 3 times a day (TID), 140 mg TID and 280 mg TID.
  Cisplatin will be administered intravenously at a dose of 40 mg/m^2 on Days 1, 8, 15, 22, 29, 36, and 43 of the 7-week concurrent treatment course.
  The prescribed radiotherapy dose will be 70 Gray (Gy) in 2 Gy once-daily fraction size (total of 35 fractions) over the 7-week concurrent treatment course. The initial target volume encompassing the gross and subclinical disease sites will receive 2.0 Gy per fraction, 5 fractions per week.
  Interventions: Drug: oral rigosertib; Drug: cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: oral rigosertib
  Other Names: ON 01910.Na; rigosertib sodium
Drug: cisplatin
Radiation: Radiotherapy

SUMMARY:
The working hypothesis is that oral rigosertib treatment when added to platinum-based Chemoradiotherapy (CRT) will improve progression-free survival for first-line patients with intermediate- or high-risk human papillomavirus negative positive (HPV (+)) Head and Neck Squamous Cell Carcinoma. This study will determine the highest safe dose of oral rigosertib that can be used with cisplatin and CRT. This study will also record any side effects that may occur and measure tumor sizes and how long patients live.

DETAILED DESCRIPTION:
This is a multicenter, dose-escalating study of oral rigosertib administered with concurrent cisplatin and Radiotherapy in patients with intermediate- and high-risk Head and Neck Squamous Cell Carcinoma.

Three rigosertib escalating cohorts (up to 6 patients per cohort) will be sequentially evaluated: 70 mg 3 times a day (TID), 140 mg TID and 280 mg TID. The total treatment course will be 8 weeks: 1 week of oral rigosertib alone (70 mg TID, 140 mg TID or 280 mg TID) followed by 7 weeks of concurrent administration of rigosertib, cisplatin and radiation therapy.

After completion of treatment, patients will be followed for up to 36 months to document Progression-free Survival and Overall Survival.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of Squamous Cell Carcinoma of the oropharynx (tonsil, base of tongue, soft palate, or oropharyngeal wall), hypopharynx, or larynx.
2. Patient is an appropriate candidate for definitive chemoradiotherapy.
3. Intermediate-risk Head and Neck Squamous Cell Carcinoma (HNSCC), defined as follows:

   1. Clinical stage T2-4, N2a-N3 or T3-4, N0-N3
   2. P16 (+) by immunohistochemistry (IHC) or HPV (+) by in situ hybridization (ISH)
   3. Smoking status of ≥ 10 pack-years, or < 10 pack-years and T4 or N2c-N3.
4. If not intermediate-risk HNSCC, is high-risk HNSCC, defined as follows:

   1. Clinical stage T2-4, N2a-N3 or T3-4, N0-N3.
   2. P16 (-) by IHC or HPV (-) by ISH.
5. No evidence of distant metastases.
6. Clinically or radiographically evident measurable disease (as defined by RECIST v 1.1) at the primary site or nodal stations.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Adequate hematologic function as defined by absolute neutrophil count (ANC) ≥ 1800/μL; platelet (PLT) ≥ 100,000/μL; Hgb ≥ 8.0 g/dL.
9. Adequate renal function, as defined by serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min.
10. Adequate liver function as defined by total bilirubin ≤ 1.5 x ULN; aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 2.5 x ULN; and prothrombin time ≤ 1.5 x ULN, unless receiving therapeutic anticoagulation.
11. Ability to understand the nature of the study and any hazards of study participation, to communicate satisfactorily with the Investigator, and to follow the requirements of the entire protocol.
12. Willingness to adhere to the prohibitions and restrictions specified in this protocol.
13. The patient must sign an informed consent form (ICF) indicating that s/he understands the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

1. Gross total excision of the primary and nodal disease.
2. Prior treatment with IV or oral rigosertib.
3. Prior chemotherapy for the study HNSCC cancer.
4. Prior radiotherapy to the region of the study HNSCC cancer or adjacent anatomical sites, or to > 25% of marrow-bearing area.
5. Synchronous malignancies.
6. Prior invasive malignancy unless the patient is disease-free for a minimum of 3 years; however, patients with prior non-melanoma skin cancer, cervical intraepithelial neoplasia (CIN), or prostate cancer with undetectable prostate-specific antigen (PSA) may be enrolled.
7. Severe, active comorbidity.
8. Known infection with human immunodeficiency virus (HIV).
9. Any uncontrolled condition that, in the opinion of the Investigator, could affect the subject's participation in the study.
10. Major surgery within 3 weeks of enrollment or major surgery without full recovery.
11. Ascites requiring active medical management, including paracentesis.
12. Hyponatremia (defined as serum sodium < 130 milliequivalent mEq/L) or conditions that may predispose patients to hyponatremia.
13. Uncontrolled hypertension, defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 110 mmHg, despite treatment with 2 antihypertensive agents.
14. New onset of seizures within 3 months prior to enrollment, or poorly controlled seizures.
15. Female patients who are pregnant or lactating.
16. Female patients of childbearing potential and male patients with partners of childbearing potential who are unwilling to follow strict contraception requirements.
17. Female patients of childbearing potential who do not have a negative blood or urine pregnancy test at Screening.
18. History of allergic reactions attributed to compounds of similar chemical or biologic composition to rigosertib.
19. Prior therapy with a phosphatidyl-inositol 3 kinase (PI3K), Akt or mammalian target of rapamycin (mTOR) inhibitor.
20. Any other investigational agent or chemotherapy, radiotherapy, or immunotherapy within 4 weeks of enrollment.
21. Psychiatric illness/social situations that would limit the patient's ability to tolerate and/or comply with study requirements, or inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who experience dose limiting toxicities | Up to 12 weeks
  The primary objective of the study is to determine the maximum tolerated dose (MTD) of oral rigosertib when administered with platinum-based chemoradiotherapy to patients with intermediate- and high-risk Head and Neck Squamous Cell Carcinoma. The MTD is defined as the dose level immediately below that at which 2 or more patients experience a dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Number of patients who experience adverse events | Up to 14 weeks
Number of patients who achieve a complete response or a partial response | Up to 3 years
  Complete response (CR) and Partial response (PR) are evaluated according to "New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1)." European Journal of Cancer, 45 (2009) 228-247.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Jimeno, MD, PhD, Study Chair — University of Colorado, Denver
Locations (4):
- United States (4):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Christiana Care Health Services, Newark, Delaware
  - Montefiore Medical Center, The Bronx, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.